CLINICAL TRIAL: NCT02791763
Title: A 52-week, Phase III, Open-label, Multi-center Study to Evaluate Efficacy and Safety of GSK1278863 in Japanese Non-dialysis and Peritoneal Dialysis Subjects With Anemia Associated With Chronic Kidney Disease
Brief Title: Phase III Study of GSK1278863 in Japanese Non-dialysis (ND) and Peritoneal Dialysis (PD) Subjects With Renal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201753
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Anaemia
Keywords: Renal Anemia; Japanese; chronic kidney disease; Peritoneal dialysis; GSK1278863; Non-dialysis
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863; continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daprodustat in ND participants (Experimental): Eligible ND participants will receive oral daprodustat (1, 2, 4, 6, 8, 12, 18 or 24 milligrams [mg] as recommended) dose once daily for 52 weeks.
  Interventions: Drug: 1 to 4 mg tablets of GSK1278863; Drug: 6 mg GSK1278863 tablet
- Epoetin beta pegol in ND participants (Active Comparator): Eligible ND participants will receive subcutaneous (SC) epoetin beta pegol (25, 50, 75, 100, 150, 200 or 250 microgram [µg] as recommended) dose once every 2 or 4 weeks for 52 weeks.
  Interventions: Drug: Epoetin beta pegol
- Daprodustat in PD participants (Experimental): Eligible PD participants will receive oral daprodustat (1, 2, 4, 6, 8, 12, 18 or 24 mg as recommended) dose once daily for 52 weeks.
  Interventions: Drug: 1 to 4 mg tablets of GSK1278863; Drug: 6 mg GSK1278863 tablet

INTERVENTIONS:
Drug: 1 to 4 mg tablets of GSK1278863 — 7.0 millimeters (mm) round, standard biconvex, white film coated tablets containing 1 mg, 2 mg, or 4 mg of GSK1278863 as active ingredient, to be orally administered once daily.
  Arms: Daprodustat in ND participants; Daprodustat in PD participants
Drug: 6 mg GSK1278863 tablet — 9.0 mm round, standard biconvex, white film coated tablets containing 6 mg of GSK1278863 as active ingredient, to be orally administered once daily.
  Arms: Daprodustat in ND participants; Daprodustat in PD participants
Drug: Epoetin beta pegol — An injectable formulation containing 25 micrograms µg, 50 µg, 75 µg, 100 µg, 150 µg, 200 µg, or 250 µg of epoetin beta pegol per syringe (0.3 mL), supplied as a glass syringe prefilled with epoetin beta pegol solution (clear colorless to pale yellow). Epoetin beta pegol will be subcutaneously administered once every 2 or 4 weeks.
  Arms: Epoetin beta pegol in ND participants

SUMMARY:
This is a Phase III, open-label, active-controlled, parallel-group, multi-center study to compare the efficacy and safety of GSK1278863 administered for 52 weeks versus epoetin beta pegol in approximately 286 Japanese ND and 50 PD subjects with renal anemia. The study will consist of three cohorts. Cohort 1 and Cohort 3 will consist of ND subjects (Erythropoiesis-Stimulating Agent [ESA] users and ESA non-users) randomized to receive GSK1278863 or epoetin beta pegol in a ratio of 1:1. PD subjects will be enrolled into Cohort 2 and will receive GSK1278863. This study consists of a 4-week screening phase, a 52-week treatment phase (including primary efficacy evaluation period [Weeks 40 to 52]), and a 4-week follow-up phase following the treatment phase. The primary objective of this study is to demonstrate non-inferiority of GSK1278863 to epoetin beta pegol based on mean hemoglobin (Hgb) during the primary efficacy evaluation period in ND subjects. ESA non-users from Cohort 1 will be excluded from the primary efficacy analysis. Study results will be used as pivotal study data for an NDA submitted for GSK1278863 for the treatment of renal anemia in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Age (at the time of informed consent): >=20 years of age
* Screening verification only: Stage of chronic kidney disease (CKD) (ND subjects only): CKD stages 3, 4, and 5 defined by estimated glomerular filtration rate (eGFR) using the Japanese Society of Nephrology-Chronic Kidney Disease Initiatives (JSN-CKDI) formula
* Dialysis:

  * Not on dialysis for at least 12 weeks prior to screening (ND subjects)
  * On peritoneal dialysis (PD subjects)
* Use of ESA:

  * ESA non-users: Have not used ESAs for 8 weeks prior to screening
  * ESA users: Have used the same ESA for 8 weeks prior to screening. However, in the ND subjects, the dose of darbepoetin alfa or epoetin beta pegol must be stable (administered once every 4 weeks and up to one-step dose change during 8 weeks prior to screening).
* Hgb: Determined at the site using an Hgb analyzer

  * ESA non-users: >=8.0 g/dL and <11.0 g/dL
  * ESA users: >=9.0 g/dL and <=13.0 g/dL
* Iron parameters: Ferritin >100 nanograms per milliliters (ng/mL) or transferrin saturation (TSAT) >20% (screening verification only)
* Gender (screening verification only): Female or male. Females: Not pregnant [demonstrated to be negative for human chorionic gonadotropin (hCG) in urine or serum], not breast-feeding, and meet at least one of the following:

  1. Females of non-childbearing potential are defined as follows:

     * Pre-menopausal with at least one of the following and no plans to utilize assisted reproductive techniques (e.g., in vitro fertilization or donor embryo transfer):
     * History of bilateral tubal ligation or salpingectomy
     * History of hysteroscopic tubal occlusion and postoperatively documented bilateral tubal obstruction
     * History of hysterectomy
     * History of bilateral oophorectomy
     * Postmenopausal defined as: females 60 years of age or older or ; In females <60 years of age, 12 months of spontaneous amenorrhea (in questionable cases a blood sample with postmenopausal follicle stimulating hormone [FSH] and estradiol concentrations is confirmatory [specified reference ranges]). Females on hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use one of the most effective contraception methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
  2. Females of childbearing potential must agree to comply with one of the contraception methods listed as requirements in "GSK Listing of Most Effective Contraceptive Methods for Females of Childbearing Potential" from 28 days prior to the first dose of study medication until the completion of the follow-up visit (for subjects randomized to the GSK1278863 group) or 7 weeks after the last dose of study treatment (for subjects randomized to the Epoetin beta pegol group).
* Informed consent: Written informed consent, including adherence to the requirements and conditions specified in the consent form and the protocol, must be obtained from each subject as specified in Protocol.

Exclusion Criteria:

Chronic kidney disease (CKD)-related criteria

* Dialysis

  * Cohort 1 and Cohort 3: Start or plan to initiate dialysis during the study
  * Cohort 2: Plan to stop peritoneal dialysis or start hemodialysis during the study
* Kidney transplant: Planned living-related kidney transplant during the study Anemia-related criteria
* Aplasia: History of bone-marrow hypoplasia or pure red cell aplasia
* Other causes of anemia: pernicious anemia, thalassemia, sickle cell anemia, or myelodysplastic syndromes
* Gastrointestinal (GI) bleeding: Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease OR clinically significant GI bleeding within 8 weeks prior to screening or during a period from screening to Day 1.

Cardiovascular disease-related criteria

* Myocardial infarction, acute coronary syndrome, stroke, or transient ischemic attack: Diagnosed within 8 weeks prior to screening or during a period from screening to Day 1.
* Heart failure: Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system
* QT interval corrected for heart rate (QTc) (screening verification only): QTc >500 milliseconds (msec) or QTc >530 msec in subjects with bundle branch block Note: QT interval corrected using the Bazett's formula (QTcB) will be used, and Electrocardiogram (ECG) can be mechanically or manually read.

Other disease-related criteria

* Liver disease (if any of the following occurs):

  * (Screening verification only) Alanine transaminase (ALT) >2 times upper limit of normal (ULN)
  * (Screening verification only) Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
  * Current unstable active liver or biliary disease (generally defined by the onset of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, persistent jaundice, or cirrhosis) Note: Stable liver disease (including asymptomatic gallstones, chronic hepatitis B/C, or Gilbert's syndrome) is acceptable if the subject otherwise meets entry criteria..
* Malignancy: History of malignancy within 2 years prior to screening, or currently receiving treatment for cancer, (PD subjects only) complex renal cystic >3 centimeters (cm) (II F, III or IV based on the Bosniak classification) Note (ND subjects and PD subjects): The only exception is squamous cell or basal cell carcinoma of the skin that has been definitively treated >=8 weeks before screening.
* In the opinion of the investigator, Hgb increase to the target range (11.0-13.0 g/dL) is medically risky.

Concomitant medication and other study treatment-related criteria

* Iron: Planned use of intravenous iron during the screening phase or during a period from Day 1 to Week 4 Note: Oral iron is acceptable. However, the same dose regimen must be used throughout the screening phase and from Day 1 to Week 4. Antihyperphosphatemic agents containing iron (e.g., ferric citrate hydrate) are also acceptable only if used for at least 12 weeks prior to screening. However, they must be continued throughout the screening phase from Day 1 to Week 4.
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product or epoetin beta pegol
* Drugs and supplements: Use or planned use of any prescription or non-prescription drugs or dietary supplements that are prohibited during the study period (prohibited medications: strong inducers and inhibitor of Cytochrome P450 2C8 [CYP2C8])
* Prior investigational product exposure: Use of an investigational agent within 30 days or five half lives of the investigational agent (whichever is longer)
* Prior treatment with GSK1278863: Any prior treatment with GSK1278863 for a treatment duration of >30 days

General health-related criteria

* Other conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the investigator (or subinvestigator) considers would put the subject at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- Japan (26):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shiga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokushima
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Toyama

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20805

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Nangaku M, Hamano T, Akizawa T, Tsubakihara Y, Nagai R, Okuda N, Kurata K, Nagakubo T, Jones NP, Endo Y, Cobitz AR. Daprodustat Compared with Epoetin Beta Pegol for Anemia in Japanese Patients Not on Dialysis: A 52-Week Randomized Open-Label Phase 3 Trial. Am J Nephrol. 2021;52(1):26-35. doi: 10.1159/000513103. Epub 2021 Feb 9. PMID 33561857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, active-controlled, parallel-group, multi-center study to compare the efficacy (verification of non-inferiority) and safety of GSK1278863 (daprodustat) versus epoetin beta pegol in Japanese non-dialysis (ND) participants, including an open-label non-comparative cohort of peritoneal dialysis (PD) participants.
Pre-assignment Details: A total of 56 centers, contracted in Japan, enrolled and randomized participants. A total of 455 participants were screened and 355 participants were enrolled and randomized in this study.
Groups:
- Daprodustat in ND Participants: Eligible ND participants received oral daprodustat (1, 2, 4, 6, 8, 12, 18 or 24 milligrams [mg] as recommended) dose once daily for 52 weeks.
- Epoetin Beta Pegol in ND Participants: Eligible ND participants received subcutaneous (SC) epoetin beta pegol (25, 50, 75, 100, 150, 200 or 250 microgram [µg] as recommended) dose once every 2 or 4 weeks for 52 weeks.
- Daprodustat in PD Participants: Eligible PD participants received oral daprodustat (1, 2, 4, 6, 8, 12, 18 or 24 mg as recommended) dose once daily for 52 weeks.
Period: Overall Study
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants | Daprodustat in PD Participants
Started | 149 | 150 | 56
Completed | 111 | 113 | 43
Not Completed | 38 | 37 | 13
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Needs maintenance/changes in dialysis | 16 | 19 | 5
Not completed — Cancer event | 1 | 3 | 0
Not completed — Participant had renal transplant | 3 | 0 | 0
Not completed — Met hemoglobin stopping criteria | 1 | 0 | 0
Not completed — Adverse Event | 12 | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants | Daprodustat in PD Participants | Total
Number analyzed (Participants) | 149 | 150 | 56 | 355
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (11.57) | 70.3 (9.09) | 64.4 (9.64) | 68.5 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 58 | 12 | 123
  Male | 96 | 92 | 44 | 232
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Asian- Japanese Heritage | 149 | 150 | 56 | 355

OUTCOME MEASURES:

1. Primary Outcome: Mean Hemoglobin (Hgb) During the Primary Efficacy Evaluation Period (Weeks 40 to 52) in ND Participants
Description: The mean hemoglobin during the primary efficacy evaluation period in ND participants was estimated by a statistical model using Mixed Model Repeated Measures (MMRM).
Time Frame: Weeks 40 to 52
Population: Intent to treat (ITT) Population comprised of cohort 1 participants (only erythropoiesis stimulating agent [ESA] users) and cohort 3 participants (both ESA users and ESA non-users) who were given randomization number with Hgb measurement at both Baseline and at least one scheduled visits following the Baseline.
Measure: Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Grams per deciliter (g/dL) | 11.97 (0.061) | 11.86 (0.063)
Statistical Analysis 1: Comparison: Daprodustat in ND Participants vs Epoetin Beta Pegol in ND Participants; Test type: Non-Inferiority — Non-inferiority was to be established as the lower limit of the 95% confidence interval (CI) for the treatment difference was greater than the pre-specified non-inferiority margin (-1.0 g/dL); p < .0001, Mixed model repeated measures (MMRM) — The p value on this table is one-sided and calculated for the non-inferiority assessment; Median Difference (Final Values) = 0.10, 95% CI 2-sided [-0.07 to 0.28], Standard Error of Mean 0.088 — Analysis was performed by a MMRM with covariates of treatment, Baseline Hgb, visit, treatment-by-visit interaction and Baseline-by-visit interaction

2. Secondary Outcome: Number of ND Participants With Mean Hgb in the Target Range (11.0-13.0 g/dL) During the Primary Efficacy Evaluation Period (Weeks 40 to 52)
Description: ND participants with observed mean Hgb within the target range during the primary efficacy evaluation period were summarized. Responders were defined as the participants with the mean Hgb within target range during the primary efficacy evaluation period.
Time Frame: Weeks 40 to 52
Population: Modified intent to treat (mITT) comprised of all ITT participants who had at least one Hgb measurement during the efficacy evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 88 | 87
Participants
  Responder | 81 | 80
  Non-Responder | 7 | 7
Statistical Analysis 1: Comparison: Daprodustat in ND Participants vs Epoetin Beta Pegol in ND Participants; Test type: Superiority; p = 0.4941, Regression, Logistic — The p value on this table is one-sided and calculated for the superiority assessment; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.33 to 3.04] — Analysis was performed by logistic regression with covariates of treatment, Baseline Hgb, and Baseline ESA use

3. Secondary Outcome: Percentage of ND Participants With Mean Hgb in the Target Range (11.0-13.0 g/dL) During the Primary Efficacy Evaluation Period (Weeks 40 to 52)
Description: The percentage of ND participants with observed mean Hgb within the target range during the primary efficacy evaluation period was summarized. Responders were defined as the participants with the mean Hgb within target range during the primary efficacy evaluation period.
Time Frame: Weeks 40 to 52
Population: mITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 88 | 87
Percentage of participants
  Responder | 92 | 92
  Non-Responder | 8 | 8
Statistical Analysis 1: Comparison: Daprodustat in ND Participants vs Epoetin Beta Pegol in ND Participants; Test type: Superiority; p = 0.4941, Regression, Logistic — The p value on this table is one-sided and calculated for the superiority assessment; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.33 to 3.04] — Analysis was performed by logistic regression with covariates of treatment, Baseline Hgb, and Baseline ESA use

4. Secondary Outcome: Change From Baseline in Hgb at Week 4 in ND Participants
Description: Baseline Hgb value was the value from the Day 1 visit. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data for change from Baseline in Hgb at Week 4 in ND participants is presented.
Time Frame: Baseline (Day 1) and Week 4
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 107 | 109
g/dL | 0.47 (0.878) | 0.26 (0.711)

5. Secondary Outcome: Change From Baseline in Hgb at Week 4 in PD Participants
Description: Baseline Hgb value was the value from the Day 1 visit. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data for change from Baseline in Hgb at week 4 in PD participants is presented.
Time Frame: Baseline (Day 1) and Week 4
Population: Efficacy peritoneal dialysis (PD) Population comprised of PD participants who were given randomization number with Hgb measurement at both Baseline and at least one scheduled visits following the Baseline.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
g/dL | -0.09 (0.899)

6. Secondary Outcome: Number of ND Participants by Hgb Change From Baseline Category at Week 4
Description: Baseline Hgb value was the value from the Day 1 visit. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Number of participants by Hgb change from Baseline is categorized to <=-2.0, >-2.0 and <=-1.0, >-1.0 and <=0, >0 and <=1.0, >1.0 and <=2.0, >2.0 g/dL, then is additionally categorized to within +/- 1.0 g/dL and over +/- 2.0 g/dL. Number of participants have been included in more than one category at Week 4.
Time Frame: Baseline (Day 1) and Week 4
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 107 | 109
Participants
  <=-2.0 | 1 | 2
  >-2.0 and <=-1.0 | 4 | 3
  >-1.0 and <=0 | 28 | 33
  >0 and <=1.0 | 43 | 56
  >1.0 and <=2.0 | 29 | 15
  >2.0 | 2 | 0
  within +/- 1.0 | 72 | 90
  over +/- 2.0 | 3 | 1

7. Secondary Outcome: Percentage of ND Participants by Hgb Change From Baseline Category at Week 4
Description: as for outcome 6
Time Frame: Baseline (Day 1) and Week 4
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 107 | 109
Percentage of participants
  <=-2.0 | 1 | 2
  >-2.0 and <=-1.0 | 4 | 3
  >-1.0 and <=0 | 26 | 30
  >0 and <=1.0 | 40 | 51
  >1.0 and <=2.0 | 27 | 14
  >2.0 | 2 | 0
  within +/- 1.0 | 67 | 83
  over +/- 2.0 | 3 | 1

8. Secondary Outcome: Number of PD Participants by Hgb Change From Baseline Category at Week 4
Description: as for outcome 6
Time Frame: Baseline (Day 1) and Week 4
Population: Efficacy PD Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Participants
  <=-2.0 | 0
  >-2.0 and <=-1.0 | 10
  >-1.0 and <=0 | 20
  >0 and <=1.0 | 20
  >1.0 and <=2.0 | 4
  >2.0 | 1
  within +/- 1.0 | 41
  over +/- 2.0 | 1

9. Secondary Outcome: Percentage of PD Participants by Hgb Change From Baseline Category at Week 4
Description: as for outcome 6
Time Frame: Baseline (Day 1) and Week 4
Population: Efficacy PD Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Percentage of Participants
  <=-2.0 | 0
  >-2.0 and <=-1.0 | 18
  >-1.0 and <=0 | 36
  >0 and <=1.0 | 36
  >1.0 and <=2.0 | 7
  >2.0 | 2
  within +/- 1.0 | 75
  over +/- 2.0 | 2

10. Secondary Outcome: Daprodustat Dose Level by Visit in ND Participants
Description: Daprodustat dose level at each assessment visit for ND participants is presented using 25th percentile (P25), median, and 75th percentile (P75).
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44 and 48
Population: ITT Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Milligrams per day (mg/day)
Arm/Group | Daprodustat in ND Participants
Number analyzed (Participants) | 108
Milligrams per day (mg/day)
  Day 1, n=108 | 4.0 [2.0 to 4.0]
  Week 4, n=106: number analyzed (Participants) | 106
  Week 4, n=106 | 4.0 [2.0 to 6.0]
  Week 8, n=106: number analyzed (Participants) | 106
  Week 8, n=106 | 4.0 [2.0 to 6.0]
  Week 12, n=106: number analyzed (Participants) | 106
  Week 12, n=106 | 4.0 [2.0 to 6.0]
  Week 16, n=103: number analyzed (Participants) | 103
  Week 16, n=103 | 4.0 [2.0 to 6.0]
  Week 20, n=100: number analyzed (Participants) | 100
  Week 20, n=100 | 4.0 [2.0 to 8.0]
  Week 24, n=96: number analyzed (Participants) | 96
  Week 24, n=96 | 4.0 [2.0 to 8.0]
  Week 28, n=94: number analyzed (Participants) | 94
  Week 28, n=94 | 4.0 [2.0 to 8.0]
  Week 32, n=92: number analyzed (Participants) | 92
  Week 32, n=92 | 4.0 [2.0 to 6.0]
  Week 36, n=89: number analyzed (Participants) | 89
  Week 36, n=89 | 4.0 [2.0 to 6.0]
  Week 40, n=88: number analyzed (Participants) | 88
  Week 40, n=88 | 4.0 [2.0 to 6.0]
  Week 44, n=88: number analyzed (Participants) | 88
  Week 44, n=88 | 4.0 [2.0 to 7.0]
  Week 48, n=87: number analyzed (Participants) | 87
  Week 48, n=87 | 4.0 [2.0 to 6.0]

11. Secondary Outcome: Epoetin Beta Pegol Dose Level by Visit in ND Participants
Description: Dose of epoetin beta pegol at a scheduled visit was converted to dose per 4 weeks when the dose frequency was every 2 weeks. Epoetin beta pegol dose level at each assessment visit for ND participants is presented using 25th percentile (P25), median, and 75th percentile (P75).
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44 and 48
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Micrograms per 4 weeks
Arm/Group | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 109
Micrograms per 4 weeks
  Day 1, n=109 | 50.0 [50.0 to 50.0]
  Week 4, n=109 | 75.0 [50.0 to 100.0]
  Week 8, n=107: number analyzed (Participants) | 107
  Week 8, n=107 | 100.0 [50.0 to 100.0]
  Week 12, n=105: number analyzed (Participants) | 105
  Week 12, n=105 | 100.0 [50.0 to 150.0]
  Week 16, n=104: number analyzed (Participants) | 104
  Week 16, n=104 | 75.0 [25.0 to 150.0]
  Week 20, n=100: number analyzed (Participants) | 100
  Week 20, n=100 | 75.0 [50.0 to 150.0]
  Week 24, n=97: number analyzed (Participants) | 97
  Week 24, n=97 | 75.0 [50.0 to 150.0]
  Week 28, n=92: number analyzed (Participants) | 92
  Week 28, n=92 | 75.0 [50.0 to 150.0]
  Week 32, n=90: number analyzed (Participants) | 90
  Week 32, n=90 | 75.0 [50.0 to 150.0]
  Week 36, n=88: number analyzed (Participants) | 88
  Week 36, n=88 | 75.0 [75.0 to 150.0]
  Week 40, n=87: number analyzed (Participants) | 87
  Week 40, n=87 | 75.0 [50.0 to 150.0]
  Week 44, n=84: number analyzed (Participants) | 84
  Week 44, n=84 | 100.0 [62.5 to 150.0]
  Week 48, n=82: number analyzed (Participants) | 82
  Week 48, n=82 | 100.0 [75.0 to 150.0]

12. Secondary Outcome: Daprodustat Dose Level by Visit in PD Participants
Description: Daprodustat dose level at each assessment visit for PD participants is presented using 25th percentile (P25), median, and 75th percentile (P75).
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44 and 48
Population: Efficacy PD Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Median (Inter-Quartile Range); unit: mg/day
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
mg/day
  Day 1, n=55 | 4.0 [4.0 to 4.0]
  Week 4, n=55 | 6.0 [4.0 to 6.0]
  Week 8, n=52: number analyzed (Participants) | 52
  Week 8, n=52 | 6.0 [4.0 to 8.0]
  Week 12, n=52: number analyzed (Participants) | 52
  Week 12, n=52 | 6.0 [4.0 to 8.0]
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | 6.0 [4.0 to 8.0]
  Week 20, n=50: number analyzed (Participants) | 50
  Week 20, n=50 | 6.0 [4.0 to 12.0]
  Week 24, n=48: number analyzed (Participants) | 48
  Week 24, n=48 | 8.0 [4.0 to 12.0]
  Week 28, n=45: number analyzed (Participants) | 45
  Week 28, n=45 | 8.0 [4.0 to 8.0]
  Week 32, n=45: number analyzed (Participants) | 45
  Week 32, n=45 | 6.0 [4.0 to 8.0]
  Week 36, n=45: number analyzed (Participants) | 45
  Week 36, n=45 | 8.0 [4.0 to 12.0]
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | 6.0 [2.0 to 8.0]
  Week 44, n=43: number analyzed (Participants) | 43
  Week 44, n=43 | 6.0 [2.0 to 8.0]
  Week 48, n=43: number analyzed (Participants) | 43
  Week 48, n=43 | 6.0 [2.0 to 8.0]

13. Secondary Outcome: Duration of Treatment Interruption Due to Hgb >13 g/dL in ND Participants
Description: The duration (in days) of treatment interruption due to Hgb >13 g/dL per participant was summarized descriptively on participants with a period of treatment interruption due to Hgb >13 g/dL.
Time Frame: Up to Week 52
Population: ITT Population. Only those participants who had Hgb > 13.0 g/dL of Hemocue were included in analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 42 | 39
Days | 28.0 [14 to 111] | 28.0 [26 to 113]

14. Secondary Outcome: Duration of Treatment Interruption Due to Hgb >13 g/dL in PD Participants
Description: as for outcome 13
Time Frame: Up to Week 52
Population: Efficacy PD Population. Only those participants who had Hgb > 13.0 g/dL of Hemocue were included in analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 23
Days | 28.0 [19 to 168]

15. Secondary Outcome: Number of Dose Adjustments in ND Participants
Description: Number of dose adjustments in ND participants is presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Median (Full Range); unit: Number of dose adjustments
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Number of dose adjustments | 5.0 [0 to 9] | 6.0 [1 to 10]

16. Secondary Outcome: Number of Dose Adjustments in PD Participants
Description: Number of dose adjustments in PD participants is presented.
Time Frame: Up to Week 52
Population: Efficacy PD Population
Measure: Median (Full Range); unit: Number of dose adjustments
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Number of dose adjustments | 5.0 [0 to 11]

17. Secondary Outcome: Hgb Values at Each Assessment Visit in ND Participants
Description: Hgb values at each assessment visit for ND participants is presented.
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
g/dL
  Day 1, n=108,109 | 10.48 (1.140) | 10.68 (1.066)
  Week 4, n=107,109: number analyzed (Participants) | 107 | 109
  Week 4, n=107,109 | 10.95 (1.122) | 10.94 (1.024)
  Week 8, n=107,109: number analyzed (Participants) | 107 | 109
  Week 8, n=107,109 | 11.19 (1.092) | 11.34 (0.905)
  Week 12, n=106,107: number analyzed (Participants) | 106 | 107
  Week 12, n=106,107 | 11.51 (1.024) | 11.84 (0.880)
  Week 16, n=104,105: number analyzed (Participants) | 104 | 105
  Week 16, n=104,105 | 11.90 (1.091) | 12.07 (1.073)
  Week 20, n=102,103: number analyzed (Participants) | 102 | 103
  Week 20, n=102,103 | 11.84 (0.909) | 11.96 (0.820)
  Week 24, n=99,99: number analyzed (Participants) | 99 | 99
  Week 24, n=99,99 | 11.87 (0.740) | 11.80 (0.855)
  Week 28, n=96,93: number analyzed (Participants) | 96 | 93
  Week 28, n=96,93 | 11.98 (0.845) | 11.83 (0.859)
  Week 32, n=92,90: number analyzed (Participants) | 92 | 90
  Week 32, n=92,90 | 12.03 (0.785) | 11.80 (0.875)
  Week 36, n=92,88: number analyzed (Participants) | 92 | 88
  Week 36, n=92,88 | 11.93 (0.730) | 11.81 (0.810)
  Week 40, n=88,87: number analyzed (Participants) | 88 | 87
  Week 40, n=88,87 | 11.88 (0.735) | 12.00 (0.857)
  Week 44, n=88,86: number analyzed (Participants) | 88 | 86
  Week 44, n=88,86 | 11.87 (0.868) | 11.75 (0.763)
  Week 48, n=87,83: number analyzed (Participants) | 87 | 83
  Week 48, n=87,83 | 12.05 (0.896) | 11.80 (0.904)
  Week 52, n=87,81: number analyzed (Participants) | 87 | 81
  Week 52, n=87,81 | 12.01 (1.003) | 11.99 (0.930)

18. Secondary Outcome: Hgb Values at Each Assessment Visit in PD Participants
Description: Hgb values at each assessment visit for PD participants is presented.
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
g/dL
  Day 1, n=55 | 10.85 (0.964)
  Week 4, n=55 | 10.77 (1.239)
  Week 8, n=54: number analyzed (Participants) | 54
  Week 8, n=54 | 10.83 (1.259)
  Week 12, n=52: number analyzed (Participants) | 52
  Week 12, n=52 | 11.36 (1.097)
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | 11.42 (1.079)
  Week 20, n=50: number analyzed (Participants) | 50
  Week 20, n=50 | 11.54 (0.807)
  Week 24, n=49: number analyzed (Participants) | 49
  Week 24, n=49 | 11.69 (0.816)
  Week 28, n=48: number analyzed (Participants) | 48
  Week 28, n=48 | 11.95 (1.038)
  Week 32, n=45: number analyzed (Participants) | 45
  Week 32, n=45 | 12.07 (0.890)
  Week 36, n=45: number analyzed (Participants) | 45
  Week 36, n=45 | 11.90 (0.839)
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | 12.12 (0.795)
  Week 44, n=43: number analyzed (Participants) | 43
  Week 44, n=43 | 11.92 (0.824)
  Week 48, n=43: number analyzed (Participants) | 43
  Week 48, n=43 | 12.10 (0.774)
  Week 52, n=43: number analyzed (Participants) | 43
  Week 52, n=43 | 12.12 (0.699)

19. Secondary Outcome: Change From Baseline in Hgb Values at Each Assessment Visit in ND Participants
Description: Baseline Hgb value was the value from the Day 1 visit. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data for change from Baseline in Hgb values at each assessment visit in ND participants is presented.
Time Frame: Baseline (Day 1), Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 107 | 109
g/dL
  Week 4, n=107,109 | 0.47 (0.878) | 0.26 (0.711)
  Week 8, n=107,109 | 0.71 (1.122) | 0.66 (1.109)
  Week 12, n=106,107: number analyzed (Participants) | 106 | 107
  Week 12, n=106,107 | 1.04 (1.352) | 1.18 (1.384)
  Week 16, n=104,105: number analyzed (Participants) | 104 | 105
  Week 16, n=104,105 | 1.45 (1.376) | 1.40 (1.495)
  Week 20, n=102,103: number analyzed (Participants) | 102 | 103
  Week 20, n=102,103 | 1.39 (1.330) | 1.26 (1.336)
  Week 24, n=99,99: number analyzed (Participants) | 99 | 99
  Week 24, n=99,99 | 1.41 (1.346) | 1.10 (1.295)
  Week 28, n=96,93: number analyzed (Participants) | 96 | 93
  Week 28, n=96,93 | 1.54 (1.375) | 1.08 (1.151)
  Week 32, n=92,90: number analyzed (Participants) | 92 | 90
  Week 32, n=92,90 | 1.60 (1.371) | 1.04 (1.299)
  Week 36, n=92,88: number analyzed (Participants) | 92 | 88
  Week 36, n=92,88 | 1.49 (1.265) | 1.04 (1.294)
  Week 40, n=88,87: number analyzed (Participants) | 88 | 87
  Week 40, n=88,87 | 1.44 (1.371) | 1.26 (1.304)
  Week 44, n=88,86: number analyzed (Participants) | 88 | 86
  Week 44, n=88,86 | 1.43 (1.435) | 1.01 (1.131)
  Week 48, n=87,83: number analyzed (Participants) | 87 | 83
  Week 48, n=87,83 | 1.61 (1.350) | 1.03 (1.172)
  Week 52, n=87,81: number analyzed (Participants) | 87 | 81
  Week 52, n=87,81 | 1.56 (1.527) | 1.21 (1.432)

20. Secondary Outcome: Change From Baseline in Hgb Values at Each Assessment Visit in PD Participants
Description: Baseline Hgb value was the value from the Day 1 visit. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data for change from Baseline in Hgb values at each assessment visit in PD participants is presented.
Time Frame: Baseline (Day 1), Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
g/dL
  Week 4, n=55 | -0.09 (0.899)
  Week 8, n=54: number analyzed (Participants) | 54
  Week 8, n=54 | -0.06 (1.127)
  Week 12, n=52: number analyzed (Participants) | 52
  Week 12, n=52 | 0.44 (1.173)
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | 0.52 (1.295)
  Week 20, n=50: number analyzed (Participants) | 50
  Week 20, n=50 | 0.63 (1.158)
  Week 24, n=49: number analyzed (Participants) | 49
  Week 24, n=49 | 0.74 (1.182)
  Week 28, n=48: number analyzed (Participants) | 48
  Week 28, n=48 | 1.00 (1.317)
  Week 32, n=45: number analyzed (Participants) | 45
  Week 32, n=45 | 1.13 (1.192)
  Week 36, n=45: number analyzed (Participants) | 45
  Week 36, n=45 | 0.95 (1.106)
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | 1.13 (1.227)
  Week 44, n=43: number analyzed (Participants) | 43
  Week 44, n=43 | 0.90 (1.093)
  Week 48, n=43: number analyzed (Participants) | 43
  Week 48, n=43 | 1.08 (1.248)
  Week 52, n=43: number analyzed (Participants) | 43
  Week 52, n=43 | 1.10 (1.226)

21. Secondary Outcome: Number of ND Participants Who Had Hgb Level Within the Target Range (11.0-13.0 g/dL) at Each Assessment Visit
Description: Number of ND participants with Hgb level within the target range (11.0 to 13.0 g/dL) are summarized at each assessment visit.
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Participants
  Day 1, n=108,109 | 29 | 36
  Week 4, n=107,109: number analyzed (Participants) | 107 | 109
  Week 4, n=107,109 | 43 | 48
  Week 8, n=107,109: number analyzed (Participants) | 107 | 109
  Week 8, n=107,109 | 64 | 73
  Week 12, n=106,107: number analyzed (Participants) | 106 | 107
  Week 12, n=106,107 | 78 | 85
  Week 16, n=104,105: number analyzed (Participants) | 104 | 105
  Week 16, n=104,105 | 84 | 80
  Week 20, n=102,103: number analyzed (Participants) | 102 | 103
  Week 20, n=102,103 | 88 | 85
  Week 24, n=99,99: number analyzed (Participants) | 99 | 99
  Week 24, n=99,99 | 86 | 85
  Week 28, n=96,93: number analyzed (Participants) | 96 | 93
  Week 28, n=96,93 | 77 | 73
  Week 32, n=92,90: number analyzed (Participants) | 92 | 90
  Week 32, n=92,90 | 79 | 67
  Week 36, n=92,88: number analyzed (Participants) | 92 | 88
  Week 36, n=92,88 | 79 | 70
  Week 40, n=88,87: number analyzed (Participants) | 88 | 87
  Week 40, n=88,87 | 78 | 72
  Week 44, n=88,86: number analyzed (Participants) | 88 | 86
  Week 44, n=88,86 | 71 | 68
  Week 48, n=87,83: number analyzed (Participants) | 87 | 83
  Week 48, n=87,83 | 75 | 62
  Week 52, n=87,81: number analyzed (Participants) | 87 | 81
  Week 52, n=87,81 | 67 | 59

22. Secondary Outcome: Percentage of ND Participants Who Had Hgb Level Within the Target Range (11.0-13.0 g/dL) at Each Assessment Visit
Description: Percentage of ND participants with Hgb level within the target range (11.0 to 13.0 g/dL) are summarized at each assessment visit.
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Percentage of Participants
  Day 1, n=108,109 | 27 | 33
  Week 4, n=107,109: number analyzed (Participants) | 107 | 109
  Week 4, n=107,109 | 40 | 44
  Week 8, n=107,109: number analyzed (Participants) | 107 | 109
  Week 8, n=107,109 | 60 | 67
  Week 12, n=106,107: number analyzed (Participants) | 106 | 107
  Week 12, n=106,107 | 74 | 79
  Week 16, n=104,105: number analyzed (Participants) | 104 | 105
  Week 16, n=104,105 | 81 | 76
  Week 20, n=102,103: number analyzed (Participants) | 102 | 103
  Week 20, n=102,103 | 86 | 83
  Week 24, n=99,99: number analyzed (Participants) | 99 | 99
  Week 24, n=99,99 | 87 | 86
  Week 28, n=96,93: number analyzed (Participants) | 96 | 93
  Week 28, n=96,93 | 80 | 78
  Week 32, n=92,90: number analyzed (Participants) | 92 | 90
  Week 32, n=92,90 | 86 | 74
  Week 36, n=92,88: number analyzed (Participants) | 92 | 88
  Week 36, n=92,88 | 86 | 80
  Week 40, n=88,87: number analyzed (Participants) | 88 | 87
  Week 40, n=88,87 | 89 | 83
  Week 44, n=88,86: number analyzed (Participants) | 88 | 86
  Week 44, n=88,86 | 81 | 79
  Week 48, n=87,83: number analyzed (Participants) | 87 | 83
  Week 48, n=87,83 | 86 | 75
  Week 52, n=87,81: number analyzed (Participants) | 87 | 81
  Week 52, n=87,81 | 77 | 73

23. Secondary Outcome: Number of PD Participants Who Had Hgb Level Within the Target Range (11.0-13.0 g/dL) at Each Assessment Visit
Description: Number of PD participants with Hgb level within the target range (11.0 to 13.0 g/dL) are summarized at each assessment visit.
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Participants
  Day 1, n=55 | 28
  Week 4, n=55 | 25
  Week 8, n=54: number analyzed (Participants) | 54
  Week 8, n=54 | 26
  Week 12, n=52: number analyzed (Participants) | 52
  Week 12, n=52 | 32
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | 32
  Week 20, n=50: number analyzed (Participants) | 50
  Week 20, n=50 | 38
  Week 24, n=49: number analyzed (Participants) | 49
  Week 24, n=49 | 36
  Week 28, n=48: number analyzed (Participants) | 48
  Week 28, n=48 | 39
  Week 32, n=45: number analyzed (Participants) | 45
  Week 32, n=45 | 34
  Week 36, n=45: number analyzed (Participants) | 45
  Week 36, n=45 | 36
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | 34
  Week 44, n=43: number analyzed (Participants) | 43
  Week 44, n=43 | 33
  Week 48, n=43: number analyzed (Participants) | 43
  Week 48, n=43 | 36
  Week 52, n=43: number analyzed (Participants) | 43
  Week 52, n=43 | 38

24. Secondary Outcome: Percentage of PD Participants Who Had Hgb Level Within the Target Range (11.0-13.0 g/dL) at Each Assessment Visit
Description: Percentage of PD participants with Hgb level within the target range (11.0 to 13.0 g/dL) are summarized at each assessment visit.
Time Frame: Day 1, Weeks 4,8,12,16,20,24,28,32,36,40,44,48 and Week 52
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Percentage of Participants
  Day 1, n=55 | 51
  Week 4, n=55 | 45
  Week 8, n=54: number analyzed (Participants) | 54
  Week 8, n=54 | 48
  Week 12, n=52: number analyzed (Participants) | 52
  Week 12, n=52 | 62
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | 63
  Week 20, n=50: number analyzed (Participants) | 50
  Week 20, n=50 | 76
  Week 24, n=49: number analyzed (Participants) | 49
  Week 24, n=49 | 73
  Week 28, n=48: number analyzed (Participants) | 48
  Week 28, n=48 | 81
  Week 32, n=45: number analyzed (Participants) | 45
  Week 32, n=45 | 76
  Week 36, n=45: number analyzed (Participants) | 45
  Week 36, n=45 | 80
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | 77
  Week 44, n=43: number analyzed (Participants) | 43
  Week 44, n=43 | 77
  Week 48, n=43: number analyzed (Participants) | 43
  Week 48, n=43 | 84
  Week 52, n=43: number analyzed (Participants) | 43
  Week 52, n=43 | 88

25. Secondary Outcome: Percentage of Time With Hgb Within the Target Range (11.0 to 13.0 g/dL) During the Primary Efficacy Evaluation Period (Weeks 40 to 52) in ND Participants
Description: Mean percentage of time with Hgb within the target range (11.0 to 13.0 g/dL) is summarized during the primary efficacy evaluation period (Weeks 40 to 52).
Time Frame: Weeks 40 to 52
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 88 | 87
Percentage of time | 85.44 (22.473) | 80.57 (25.973)

26. Secondary Outcome: Percentage of Time With Hgb Within the Target Range (11.0 to 13.0 g/dL) During the Primary Efficacy Evaluation Period (Weeks 40 to 52) in PD Participants
Description: as for outcome 25
Time Frame: Weeks 40 to 52
Population: Efficacy PD Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 44
Percentage of time | 85.73 (19.974)

27. Secondary Outcome: Time to Reach the Lower Target Hgb Level (11.0 g/dL) in ND Participants
Description: The time (in days) to reach the lower target Hgb level (11.0 g/dL) was summarized using 25th percentile (P25), median, and 75th percentile (P75) by Kaplan-Meier method. Participants who did not reach the lower Hgb target were considered as censored cases. Participants who were randomized as Hgb >= 11.0 g/dL were excluded in this summary.
Time Frame: Up to week 52
Population: ITT Population. Only those participants who experienced this event were included in analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 76 | 75
Days | 58.0 [29.0 to 87.0] | 57.0 [29.0 to 85.0]

28. Secondary Outcome: Time to Reach the Lower Target Hgb Level (11.0 g/dL) in PD Participants
Description: as for outcome 27
Time Frame: Up to week 52
Population: Efficacy PD Population. Only those participants who experienced this event were included in analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 27
Days | 84.0 [29.0 to 141.0]

29. Secondary Outcome: Number of ND Participants Who Had an Hgb Level of Less Than 7.5 g/dL
Description: Number of ND participants who had an Hgb level of less than 7.5 g/dL is presented.
Time Frame: Up to week 52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Participants | 1 | 0

30. Secondary Outcome: Percentage of ND Participants Who Had an Hgb Level of Less Than 7.5 g/dL
Description: Percentage of ND participants who had an Hgb level of less than 7.5 g/dL is presented.
Time Frame: Up to week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Percentage of participants | 1 | 0

31. Secondary Outcome: Number of PD Participants Who Had an Hgb Level of Less Than 7.5 g/dL
Description: Number of PD participants who had an Hgb level of less than 7.5 g/dL is presented.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Participants | 0

32. Secondary Outcome: Percentage of PD Participants Who Had an Hgb Level of Less Than 7.5 g/dL
Description: Percentage of PD participants who had an Hgb level of less than 7.5 g/dL is presented.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Percentage of participants | 0

33. Secondary Outcome: Number of ND Participants Who Had an Hgb Increase of More Than 2 g/dL Over Any 4 Weeks
Description: Number of ND participants who had an Hgb increase of more than 2 g/dL over any 4 weeks is presented.
Time Frame: Up to week 52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Participants | 17 | 11

34. Secondary Outcome: Percentage of ND Participants Who Had an Hgb Increase of More Than 2 g/dL Over Any 4 Weeks
Description: Percentage of ND participants who had an Hgb increase of more than 2 g/dL over any 4 weeks is presented.
Time Frame: Up to week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Percentage of participants | 16 | 10

35. Secondary Outcome: Number of PD Participants Who Had an Hgb Increase of More Than 2 g/dL Over Any 4 Weeks
Description: Number of PD participants who had an Hgb increase of more than 2 g/dL over any 4 weeks is presented.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Participants | 11

36. Secondary Outcome: Percentage of PD Participants Who Had an Hgb Increase of More Than 2 g/dL Over Any 4 Weeks
Description: Percentage of PD participants who had an Hgb increase of more than 2 g/dL over any 4 weeks is presented.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Percentage of participants | 20

37. Secondary Outcome: Number of ND Participants Who Had an Hgb Level of More Than 13.0 g/dL
Description: Number of ND participants who had an Hgb level of more than 13.0 g/dL is presented.
Time Frame: Up to week 52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Participants | 49 | 52

38. Secondary Outcome: Percentage of ND Participants Who Had an Hgb Level of More Than 13.0 g/dL
Description: Percentage of ND participants who had an Hgb level of more than 13.0 g/dL is presented.
Time Frame: Up to week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Percentage of participants | 45 | 48

39. Secondary Outcome: Number of PD Participants Who Had an Hgb Level of More Than 13.0 g/dL
Description: Number of PD participants who had an Hgb level of more than 13.0 g/dL is presented.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Participants | 28

40. Secondary Outcome: Percentage of PD Participants Who Had an Hgb Level of More Than 13.0 g/dL
Description: Percentage of PD participants who had an Hgb level of more than 13.0 g/dL is presented.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Percentage of participants | 51

41. Secondary Outcome: Number of Episodes With Hgb Level of More Than 13.0 g/dL in ND Participants
Description: Number of episodes with Hgb level of more than 13.0 g/dL in ND participants is presented.
Time Frame: Up to week 52
Population: ITT Population
Measure: Number; unit: Episodes
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Episodes | 76 | 88

42. Secondary Outcome: Number of Episodes With Hgb Level of More Than 13.0 g/dL in PD Participants
Description: Number of episodes with Hgb level of more than 13.0 g/dL in PD participants is presented.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Number; unit: Episodes
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Episodes | 43

43. Secondary Outcome: Monthly Average Dose of Oral Iron During the Treatment Period in ND Participants
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. Monthly average oral iron = Total oral iron dose (mg) / (duration in days / 30.4375 days). Monthly average dose of oral iron during the treatment period in ND participants is presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Milligrams | 837.37 (1209.100) | 747.04 (1130.767)

44. Secondary Outcome: Monthly Average Dose of Oral Iron During the Treatment Period in PD Participants
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. Monthly average oral iron = Total oral iron dose (mg) / (duration in days / 30.4375 days). Monthly average dose of oral iron during the treatment period in PD participants is presented.
Time Frame: Up to Week 52
Population: Efficacy PD Population
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Milligrams | 2468.68 (5418.767)

45. Secondary Outcome: Monthly Average Dose of Oral Iron During the Primary Efficacy Evaluation Period in ND Participants
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. Monthly average oral iron dose during the primary efficacy evaluation period (Weeks 40 to 52) = Total oral iron dose (mg) during the primary efficacy evaluation period / (duration in the period in days / 30.4375 days). Monthly average dose of oral iron during the primary efficacy evaluation period in ND participants is presented.
Time Frame: Weeks 40 to 52
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 88 | 87
Milligrams | 967.41 (1854.896) | 777.69 (1639.331)

46. Secondary Outcome: Monthly Average Dose of Oral Iron During the Primary Efficacy Evaluation Period in PD Participants
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. Monthly average oral iron dose during the primary efficacy evaluation period (Weeks 40 to 52) = Total oral iron dose (mg) during the primary efficacy evaluation period / (duration in the period in days / 30.4375 days). Monthly average dose of oral iron during the primary efficacy evaluation period in PD participants is presented.
Time Frame: Weeks 40 to 52
Population: Efficacy PD Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 44
Milligrams | 3038.67 (6239.034)

47. Secondary Outcome: Number of ND Participants Who Used Oral Iron During the Treatment Period
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. The number of ND participants who used oral iron during the treatment period were summarized.
Time Frame: Up to week 52
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Participants | 56 | 49

48. Secondary Outcome: Number of PD Participants Who Used Oral Iron During the Treatment Period
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. The number of PD participants who used oral iron during the treatment period were summarized.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Participants | 33

49. Secondary Outcome: Percentage of ND Participants Who Used Oral Iron During the Treatment Period
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. The percentage of ND participants who used oral iron during the treatment period were summarized.
Time Frame: Up to week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 108 | 109
Percentage of participants | 52 | 45

50. Secondary Outcome: Percentage of PD Participants Who Used Oral Iron During the Treatment Period
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. The percentage of PD participants who used oral iron during the treatment period were summarized.
Time Frame: Up to week 52
Population: Efficacy PD Population
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Percentage of participants | 60

51. Secondary Outcome: Number of ND Participants Who Used Oral Iron During the Primary Efficacy Evaluation Period
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. The number of ND participants who used oral iron during the primary efficacy evaluation period (Weeks 40 to 52) were summarized.
Time Frame: Weeks 40 to 52
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 88 | 87
Participants | 34 | 28

52. Secondary Outcome: Number of PD Participants Who Used Oral Iron During the Primary Efficacy Evaluation Period
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. The number of PD participants who used oral iron during the primary efficacy evaluation period (Weeks 40 to 52) were summarized.
Time Frame: Weeks 40 to 52
Population: Efficacy PD Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 44
Participants | 22

53. Secondary Outcome: Percentage of ND Participants Who Used Oral Iron During the Primary Efficacy Evaluation Period
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. The percentage of ND participants who used oral iron during the primary efficacy evaluation period (Weeks 40 to 52) were summarized.
Time Frame: Weeks 40 to 52
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 88 | 87
Percentage of participants | 39 | 32

54. Secondary Outcome: Percentage of PD Participants Who Used Oral Iron During the Primary Efficacy Evaluation Period
Description: Supplemental iron therapy were received by participants if required during treatment period. Participants who used ferric citrate were counted as oral iron use. The percentage of PD participants who used oral iron during the primary efficacy evaluation period (Weeks 40 to 52) were summarized.
Time Frame: Weeks 40 to 52
Population: Efficacy PD Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 44
Percentage of participants | 50

55. Secondary Outcome: Change From Baseline in Ferritin in ND Participants
Description: Change from Baseline in Ferritin in ND participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Adjusted mean and 95% confidence interval for change from Baseline in Ferritin is presented. For adjusted values, analysis was performed by MMRM with covariates of treatment, Baseline, visit, treatment-by-visit interaction and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: Micrograms per liter (µg/L)
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 107 | 109
Micrograms per liter (µg/L)
  Week 4, n=107,109 | -41.4 [-53.7 to -29.2] | -29.0 [-41.1 to -16.9]
  Week 16, n=104,105: number analyzed (Participants) | 104 | 105
  Week 16, n=104,105 | -83.4 [-102.8 to -64.0] | -29.3 [-48.6 to -10.0]
  Week 28, n=96,93: number analyzed (Participants) | 96 | 93
  Week 28, n=96,93 | -80.1 [-96.4 to -63.8] | -16.6 [-33.1 to -0.1]
  Week 40, n=88,87: number analyzed (Participants) | 88 | 87
  Week 40, n=88,87 | -56.3 [-79.1 to -33.4] | -16.0 [-38.9 to 6.9]
  Week 52, n=87,81: number analyzed (Participants) | 87 | 81
  Week 52, n=87,81 | -42.7 [-68.9 to -16.4] | -14.0 [-40.9 to 13.0]

56. Secondary Outcome: Change From Baseline in Ferritin in PD Participants
Description: Change from Baseline in Ferritin in PD participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Adjusted mean and 95% confidence interval for change from Baseline in Ferritin is presented. For adjusted values, analysis was performed by MMRM with covariates of Baseline, visit and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: µg/L
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
µg/L
  Week 4, n=55 | -36.4 [-49.8 to -23.1]
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | -81.8 [-103.7 to -59.9]
  Week 28, n=48: number analyzed (Participants) | 48
  Week 28, n=48 | -89.1 [-111.6 to -66.7]
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | -74.6 [-112.7 to -36.4]
  Week 52, n=43: number analyzed (Participants) | 43
  Week 52, n=43 | -63.6 [-101.0 to -26.2]

57. Secondary Outcome: Percent Change From Baseline in Transferrin Saturation (TSAT) in ND Participants
Description: Percent change from Baseline in TSAT in ND participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated as 100*(exponential [mean change on log scale]-1). Adjusted geometric mean and 95% confidence interval for percent change from Baseline in TSAT is presented. For adjusted values, analysis was performed by MMRM with covariates of treatment, Baseline, visit, treatment-by-visit interaction and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 107 | 109
Percent change
  Week 4, n=107,109 | -12.4 [-17.6 to -6.8] | -5.4 [-11.1 to 0.5]
  Week 16, n=104,105: number analyzed (Participants) | 104 | 105
  Week 16, n=104,105 | -16.3 [-21.6 to -10.6] | -0.3 [-6.6 to 6.5]
  Week 28, n=96,93: number analyzed (Participants) | 96 | 93
  Week 28, n=96,93 | -17.5 [-23.2 to -11.4] | 10.6 [2.9 to 18.9]
  Week 40, n=88,87: number analyzed (Participants) | 88 | 87
  Week 40, n=88,87 | -11.2 [-17.8 to -4.1] | 12.5 [4.1 to 21.5]
  Week 52, n=87,81: number analyzed (Participants) | 87 | 81
  Week 52, n=87,81 | -11.7 [-18.3 to -4.6] | 7.0 [-1.3 to 15.9]

58. Secondary Outcome: Percent Change From Baseline in TSAT in PD Participants
Description: Percent change from Baseline in TSAT in PD participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated as 100*(exponential [mean change on log scale]-1). Adjusted geometric mean and 95% confidence interval for percent change from Baseline in TSAT is presented. For adjusted values, analysis was performed by MMRM with covariates of Baseline, visit and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
Percent change
  Week 4, n=55 | -19.2 [-27.2 to -10.4]
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | -29.1 [-36.9 to -20.5]
  Week 28, n=48: number analyzed (Participants) | 48
  Week 28, n=48 | -22.6 [-30.4 to -14.0]
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | -19.5 [-28.3 to -9.5]
  Week 52, n=43: number analyzed (Participants) | 43
  Week 52, n=43 | -14.7 [-25.4 to -2.6]

59. Secondary Outcome: Percent Change From Baseline in Hepcidin in ND Participants
Description: Percent change from Baseline in Hepcidin in ND participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated as 100*(exponential [mean change on log scale]-1). Adjusted geometric mean and 95% confidence interval for percent change from Baseline in Hepcidin is presented. For adjusted values, analysis was performed by MMRM with covariates of treatment, Baseline, visit, treatment-by-visit interaction and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 99 | 100
Percent change
  Week 4, n=99,100 | -49.13 [-54.63 to -42.97] | -19.20 [-27.82 to -9.55]
  Week 16, n=86,99: number analyzed (Participants) | 86 | 99
  Week 16, n=86,99 | -55.67 [-61.60 to -48.82] | -3.73 [-15.95 to 10.27]
  Week 28, n=81,85: number analyzed (Participants) | 81 | 85
  Week 28, n=81,85 | -56.67 [-62.53 to -49.90] | 7.61 [-6.75 to 24.18]
  Week 40, n=76,80: number analyzed (Participants) | 76 | 80
  Week 40, n=76,80 | -47.77 [-55.10 to -39.23] | 9.54 [-5.62 to 27.12]
  Week 52, n=76,74: number analyzed (Participants) | 76 | 74
  Week 52, n=76,74 | -45.27 [-54.32 to -34.43] | 10.13 [-8.27 to 32.21]

60. Secondary Outcome: Percent Change From Baseline in Hepcidin in PD Participants
Description: Percent change from Baseline in Hepcidin in PD participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Percent change from Baseline was calculated as 100*(exponential [mean change on log scale]-1). Adjusted geometric mean and 95% confidence interval for percent change from Baseline in Hepcidin is presented. For adjusted values, analysis was performed by MMRM with covariates of Baseline, visit and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 53
Percent change
  Week 4, n=53 | -49.79 [-58.57 to -39.15]
  Week 16, n=48: number analyzed (Participants) | 48
  Week 16, n=48 | -62.59 [-69.95 to -53.42]
  Week 28, n=39: number analyzed (Participants) | 39
  Week 28, n=39 | -65.37 [-72.61 to -56.22]
  Week 40, n=39: number analyzed (Participants) | 39
  Week 40, n=39 | -67.91 [-76.10 to -56.91]
  Week 52, n=40: number analyzed (Participants) | 40
  Week 52, n=40 | -54.77 [-66.82 to -38.33]

61. Secondary Outcome: Change From Baseline in Serum Iron in ND Participants
Description: Change from Baseline in serum iron in ND participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Adjusted mean and 95% confidence interval for change from Baseline in Serum iron is presented. For adjusted values, analysis was performed by MMRM with covariates of treatment, Baseline, visit, treatment-by-visit interaction and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: Micromoles per liter (µmol/L)
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 107 | 109
Micromoles per liter (µmol/L)
  Week 4, n=107,109 | 0.5 [-0.6 to 1.5] | -0.8 [-1.8 to 0.2]
  Week 16, n=104,105: number analyzed (Participants) | 104 | 105
  Week 16, n=104,105 | 0.3 [-0.8 to 1.3] | 0.6 [-0.4 to 1.6]
  Week 28, n=96,93: number analyzed (Participants) | 96 | 93
  Week 28, n=96,93 | 0.3 [-0.8 to 1.5] | 2.0 [0.8 to 3.1]
  Week 40, n=88,87: number analyzed (Participants) | 88 | 87
  Week 40, n=88,87 | 0.9 [-0.2 to 2.1] | 1.8 [0.6 to 2.9]
  Week 52, n=87,81: number analyzed (Participants) | 87 | 81
  Week 52, n=87,81 | 0.7 [-0.4 to 1.8] | 1.1 [-0.1 to 2.2]

62. Secondary Outcome: Change From Baseline in Serum Iron in PD Participants
Description: Change from Baseline in serum iron in PD participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Adjusted mean and 95% confidence interval for change from Baseline in Serum iron is presented. For adjusted values, analysis was performed by MMRM with covariates of Baseline, visit and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: µmol/L
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
µmol/L
  Week 4, n=55 | -1.2 [-2.7 to 0.4]
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | -2.4 [-3.8 to -1.1]
  Week 28, n=48: number analyzed (Participants) | 48
  Week 28, n=48 | -1.0 [-2.5 to 0.5]
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | -0.4 [-1.9 to 1.2]
  Week 52, n=43: number analyzed (Participants) | 43
  Week 52, n=43 | 1.0 [-1.9 to 3.9]

63. Secondary Outcome: Change From Baseline in Total Iron Binding Capacity (TIBC) in ND Participants
Description: Change from Baseline in TIBC in ND participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Adjusted mean and 95% confidence interval for change from Baseline in TIBC is presented. For adjusted values, analysis was performed by MMRM with covariates of treatment, Baseline, visit, treatment-by-visit interaction and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: µmol/L
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants
Number analyzed (Participants) | 107 | 109
µmol/L
  Week 4, n=107,109 | 6.9 [6.2 to 7.7] | 0.5 [-0.2 to 1.3]
  Week 16, n=104,105: number analyzed (Participants) | 104 | 105
  Week 16, n=104,105 | 9.9 [8.7 to 11.0] | 1.9 [0.8 to 3.1]
  Week 28, n=96,93: number analyzed (Participants) | 96 | 93
  Week 28, n=96,93 | 9.9 [8.7 to 11.1] | 1.4 [0.2 to 2.6]
  Week 40, n=88,87: number analyzed (Participants) | 88 | 87
  Week 40, n=88,87 | 8.0 [6.6 to 9.4] | 0.2 [-1.2 to 1.7]
  Week 52, n=87,81: number analyzed (Participants) | 87 | 81
  Week 52, n=87,81 | 7.8 [6.3 to 9.3] | 0.1 [-1.4 to 1.7]

64. Secondary Outcome: Change From Baseline in TIBC in PD Participants
Description: Change from Baseline in TIBC in PD participants was summarized at each assessment visit. The Baseline value was the latest pre-dose assessment (Day 1 pre-dose). Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Adjusted mean and 95% confidence interval for change from Baseline in TIBC is presented. For adjusted values, analysis was performed by MMRM with covariates of Baseline, visit and Baseline-by-visit interaction.
Time Frame: Baseline (Day 1 pre-dose) and Weeks 4, 16, 28, 40 and 52
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: µmol/L
Arm/Group | Daprodustat in PD Participants
Number analyzed (Participants) | 55
µmol/L
  Week 4, n=55 | 6.9 [5.7 to 8.0]
  Week 16, n=51: number analyzed (Participants) | 51
  Week 16, n=51 | 9.5 [7.7 to 11.3]
  Week 28, n=48: number analyzed (Participants) | 48
  Week 28, n=48 | 11.0 [8.8 to 13.2]
  Week 40, n=44: number analyzed (Participants) | 44
  Week 40, n=44 | 11.0 [8.0 to 14.0]
  Week 52, n=43: number analyzed (Participants) | 43
  Week 52, n=43 | 9.6 [6.8 to 12.5]

65. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to 4 Hours (AUC[0-4]) of Daprodustat for All Dose Levels in ND and PD Participants
Description: Blood samples were collected at indicated timepoints. Pharmacokinetic (PK) parameters of Daprodustat were calculated using non-compartmental method. AUC (0-4) is presented for combined Week 12 and 24. Geometric mean and geometric coefficient of variation is presented. NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.
Time Frame: 1, 2, 3 and 4 hours post dose at Weeks 12 and 24
Population: PK Population comprised of all Daprodustat-treated participants from whom PK samples were collected and analyzed. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Groups:
- Daprodustat 1 mg: Participants received oral daprodustat tablet (1 mg) once on the day of PK sampling at Week 12 or 24.
- Daprodustat 2 mg: Participants received oral daprodustat tablet (2 mg) once on the day of PK sampling at Week 12 or 24.
- Daprodustat 4 mg: Participants received oral daprodustat tablet (4 mg) once on the day of PK sampling at Week 12 or 24.
- Daprodustat 6 mg: Participants received oral daprodustat tablet (6 mg) once on the day of PK sampling at Week 12 or 24.
- Daprodustat 8 mg: Participants received oral dose of 8 mg daprodustat (4 mg*2 tablets) once on the day of PK sampling at Week 12 or 24.
- Daprodustat 12 mg: Participants received oral dose of 12 mg of daprodustat (6 mg*2 tablets) once on the day of PK sampling at Week 12 or 24.
- Daprodustat 18 mg: Participants received oral dose of 18 mg of daprodustat (6 mg*3 tablets) once on the day of PK sampling at Week 12 or 24.
- Daprodustat 24 mg: Participants received oral dose of 24 mg of daprodustat (6 mg*4 tablets) once on the day of PK sampling at Week 12 or 24.
Arm/Group | Daprodustat 1 mg | Daprodustat 2 mg | Daprodustat 4 mg | Daprodustat 6 mg | Daprodustat 8 mg | Daprodustat 12 mg | Daprodustat 18 mg | Daprodustat 24 mg
Number analyzed (Participants) | 13 | 68 | 113 | 83 | 66 | 16 | 7 | 1
Hour*nanogram per milliliter | 35.3199 (38.4) | 63.0175 (89.8) | 101.9293 (96.5) | 152.4966 (83.2) | 167.6515 (105.9) | 190.0962 (65.9) | 435.6847 (131.7) | 404.0567 (NA) — NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.

66. Secondary Outcome: Maximum Observed Concentration (Cmax) of Daprodustat for All Dose Levels in ND and PD Participants
Description: Blood samples were collected at indicated timepoints. PK parameters of Daprodustat were calculated using non-compartmental method. Cmax is presented for combined Week 12 and 24. Geometric mean and geometric coefficient of variation is presented. NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.
Time Frame: 1, 2, 3 and 4 hours post dose at Weeks 12 and 24
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Daprodustat 1 mg | Daprodustat 2 mg | Daprodustat 4 mg | Daprodustat 6 mg | Daprodustat 8 mg | Daprodustat 12 mg | Daprodustat 18 mg | Daprodustat 24 mg
Number analyzed (Participants) | 13 | 68 | 113 | 83 | 66 | 16 | 7 | 1
Nanogram per milliliter | 17.6522 (36.5) | 35.0709 (91.2) | 58.6098 (83.2) | 81.1851 (82.6) | 91.0731 (95.4) | 94.1242 (73.3) | 197.9290 (159.6) | 226.0000 (NA) — NA indicates that the data is not available since geometric coefficient of variation could not be calculated for a single participant.

ADVERSE EVENTS:
Time Frame: On-therapy serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment up to Week 52 for both ND and PD participants.
Description: SAEs and non-serious AEs were reported treatment-wise for the Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Daprodustat in ND Participants | Epoetin Beta Pegol in ND Participants | Daprodustat in PD Participants
All-Cause Mortality (participants affected / at risk) | 1/149 | 2/150 | 0/56
Serious Adverse Events (participants affected / at risk) | 34/149 | 43/150 | 26/56
Other Adverse Events (participants affected / at risk) | 85/149 | 91/150 | 41/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat in ND Participants (N=149) | Epoetin Beta Pegol in ND Participants (N=150) | Daprodustat in PD Participants (N=56)
Renal impairment (Renal and urinary disorders) | 5 (5) | 11 (11) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 6 (6) | 8 (9) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 5 (7) | 3 (3)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 9 (12)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinocerebellar disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Steal syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat in ND Participants (N=149) | Epoetin Beta Pegol in ND Participants (N=150) | Daprodustat in PD Participants (N=56)
Nasopharyngitis (Infections and infestations) | 49 (68) | 56 (77) | 16 (23)
Influenza (Infections and infestations) | 8 (8) | 8 (9) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 9 (15)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (6)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 10 (10) | 18 (19) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 11 (13) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (14) | 7 (7) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (12) | 5 (5) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (7) | 8 (9) | 0 (0)
Blood pressure increased (Investigations) | 8 (8) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 8 (8) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
A participant in ND daprodustat/ND epoetin beta pegol/PD daprodustat had data entry error with dose level. This had an impact on outcomes of dose level and number of dose adjustment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02791763/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT02791763/SAP_001.pdf